CLINICAL TRIAL: NCT03596905
Title: A Randomized, Double-blind, Placebo-Controlled, Dose Ranging, Parallel-Group Study of the Efficacy and Safety of Plecanatide in Children 6 to <18 Years of Age With Irritable Bowel Syndrome With Constipation (IBS-C)
Brief Title: Efficacy and Safety of Plecanatide in Children 6 to <18 Years With Irritable Bowel Syndrome With Constipation (IBS-C)
Acronym: (IBS-C)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP304202-14
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Irritable Bowel Syndrome With Constipation
MeSH Terms: interventions — plecanatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- 0.5 mg plecanatide (Experimental): Plecanatide 0.5 mg Taken orally once daily for 4 weeks Group A: 6 to 11 years old
  Interventions: Drug: Plecanatide
- 1.0 mg plecanatide - Group A (Experimental): Plecanatide 1.0 mg Taken orally daily for 4 weeks Group A: 6 to 11 years old
  Interventions: Drug: Plecanatide
- 2.0 mg plecanatide (Experimental): Plecanatide 2.0 mg Taken orally daily for 4 weeks Group B: 12 to 18 Years of Age
  Interventions: Drug: Plecanatide
- 3.0 mg plecanatide (Experimental): Plecanatide 3.0 mg Taken orally daily for 4 weeks Group B: 12 to < 18 years old
  Interventions: Drug: Plecanatide
- Matching placebo - Group A (Placebo Comparator): Matching placebo Taken orally daily for 4 weeks Group A: 6 to 11 years old
  Interventions: Drug: Matching placebo
- 1.0 mg plecanatide - Group B (Experimental): Plecanatide 1.0 mg Taken orally daily for 4 weeks Group B: ≥ 12 to < 18 Years of Age
  Interventions: Drug: Plecanatide
- Matching Placebo - Group B (Placebo Comparator): Matching placebo Taken orally daily for 4 weeks Group B: 12 to < 18 years old
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Plecanatide — Taken orally daily for 4 weeks
  Other Names: Trulance
  Arms: 0.5 mg plecanatide; 1.0 mg plecanatide - Group A; 1.0 mg plecanatide - Group B; 2.0 mg plecanatide; 3.0 mg plecanatide
Drug: Matching placebo — Taken orally daily for 4 weeks
  Other Names: No other names
  Arms: Matching Placebo - Group B; Matching placebo - Group A

SUMMARY:
The goal of this clinical trial is to learn if plecanatide can improve bowel function and relieve symptoms of irritable bowel syndrome with constipation (IBS-C) in children and adolescents aged 6 to <18 years. The main questions it aims to answer are:

* Does plecanatide increase the number of spontaneous bowel movements (SBMs) compared to placebo?
* Is plecanatide safe and well tolerated in this pediatric population? Researchers will compare plecanatide at different doses to a placebo (a look-alike substance with no active drug) to see if plecanatide improves bowel function.

Participants will:

* Take plecanatide or placebo orally once daily for 4 weeks
* Complete daily symptom diaries
* Attend clinic visits for assessments and safety checks

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, dose-ranging clinical trial designed to evaluate the safety, efficacy, and pharmacokinetics of plecanatide in pediatric patients aged 6 to <18 years with irritable bowel syndrome with constipation (IBS-C). IBS-C is a condition that causes abdominal pain and infrequent, hard bowel movements.

The study includes two age cohorts:

Group A: 6 to 11 years Group B: 12 to <18 years

Participants are randomly assigned to receive one of four plecanatide doses (0.5 mg, 1.0 mg, 2.0 mg, or 3.0 mg) or placebo. All treatments were taken orally once daily for 4 weeks following a 28-day screening/baseline period. After treatment, participants were followed for 2 weeks.

The primary objective is to determine whether plecanatide increases the number of spontaneous bowel movements (SBMs) compared to placebo.

Secondary objectives include:

Time to first bowel movement after starting treatment Changes in stool consistency Changes in abdominal pain and discomfort Overall safety and tolerability of plecanatide

Safety assessments include monitoring adverse events, laboratory tests, and treatment compliance. Participants recorded daily bowel habits and symptoms in an electronic diary and attended scheduled clinic visits for evaluations.

ELIGIBILITY:
INCLUSION CRITERIA

A patient will be eligible for study participation if he or she meets all of the following criteria:

1. Male or female child or adolescent age 6 to < 18;
2. Meets ROME IV criteria for child/adolescent IBS-C defined as:

For at least 2 months before diagnosis the patient has had:

1. Abdominal pain at least 4 days per month associated with one or more of the following:

   1. Related to defecation
   2. A change in frequency of stool
   3. A change in form (appearance) of stool;
2. The pain does not resolve with resolution of the constipation (children in whom the pain resolves have functional constipation, not irritable bowel syndrome);
3. After appropriate evaluation, the symptoms cannot be fully explained by another medical condition
4. More than one-fourth (25%) of bowel movements with Bristol stool form types 1 or 2 and less than one-fourth (25%) of bowel movements with Bristol stool form types 6 or 7 on the BSFS or 4 or 5 on the mBSFS-C;

3. Patient's parent/guardian/LAR is able to voluntarily provide written, signed, and dated consent and patient is able to voluntarily provide assent as per IRB guidance; 4. Patient and patient's parent/guardian/LAR demonstrates an understanding, ability, and willingness to fully comply with protocol requirements and study procedures (e.g., acceptance of venipuncture, acceptance of urine drug screen for opiates, visit schedule, complete daily electronic diary reporting).

EXCLUSION CRITERIA

A patient will be excluded from the study if he or she meets any of the following criteria:

1. The patient has a mental age <4 years in the investigator's opinion;
2. The patient has previously been diagnosed with anorectal malformations, neurological deficits, or anatomical anomalies that would constitute a predisposition to constipation;
3. The patient currently requires iron supplements, amitriptyline, or other tricyclic antidepressants for depression, opioid-containing medications or compounds for pain, or has other conditions that require medications known to cause constipation. A patient with an onset of constipation prior to the use of these medications and who has been on a stable dose for at least 8 weeks prior to Screening might be considered eligible for this study if the investigator deems these medications do not significantly contribute to the patient's constipation. Screening of these patients needs to be approved by the medical monitor and the sponsor;
4. The patient is pregnant or lactating;
5. Females age 12 to < 18 or females age 6 to 11 of childbearing potential (defined as post menarche) who does not agree to practice one of the following medically acceptable methods of birth control throughout the study;

   * Hormonal methods such as oral, implantable, injectable, vaginal ring, or transdermal contraceptives for a minimum of 1 full cycle (based on the patient's usual menstrual cycle period) before study drug administration.
   * Total abstinence from sexual intercourse (since the last menses before study drug administration
   * Intrauterine device.
   * Double-barrier method (condoms, sponge, or diaphragm with spermicidal jellies or cream.
6. The patient follows a diet not considered normal by the investigator for the patient's age, relative to variety of food, caloric content, and quantity. The patient must have been on a stable diet for at least 30 days prior to Screening;
7. The patient's mobility or normal exercise tolerance is compromised in the investigator's opinion;
8. The patient has a history of an eating disorder;
9. The patient has clinical or laboratory signs and symptoms of significant cerebral, respiratory, renal, hepatobiliary, pancreatic, intestinal (including acute appendicitis, inflammatory bowel disease, or undiagnosed abdominal pain), endocrinologic, or infectious disease that in the investigator's judgment could interfere with study assessments or completion of the study. (Note: A patient with a history of thyroid disease may be enrolled if he or she has normal T3 and T4 at Screening. If the patient is taking medication for active thyroid disease, his or her T3 and T4 level must be within normal limits and the dose of any medication used to treat it must be stable for at least 30 days prior to Screening);
10. The patient has any other medical condition or is receiving concomitant medication or therapy that would in the investigator's opinion compromise his or her safety or compliance with the study protocol or compromise data collection;
11. The patient has a history or evidence of drug or alcohol abuse in the 12 months before Screening;
12. The patient has a hypersensitivity, allergy, or contraindication to plecanatide;
13. The patient has received any experimental drug, including linaclotide and lubiprostone, or experimental therapy within 30 days of study start;
14. The patient is unable to tolerate protocol-prescribed rescue medication (Dulcolax®), or unwilling to use it as the only laxative for the duration of the trial;
15. The patient has taken a medication considered to be a protocol-defined prohibited prior or concomitant medication or supplement as defined in section 3.3.2;
16. The patient and his or her caregiver are unable to communicate well with the study staff and comply with the study requirements (restrictions, appointments, and examination schedule). (The patient/caregiver must be able to complete required Daily BM and Symptom diary entries during the Screening/Baseline period and for the duration of the study. The patient/caregiver must also agree to provide contact information to receive daily reminders should the patient not complete the daily electronic diary entries or require password resets);
17. The patient has been screened for or participated in this or another Synergy study in the past;
18. The patient has a sibling that is currently participating or has participated in another Synergy study.

    Exclusion Criteria Based on Baseline Diary Entries
19. Patient reports having more than 1 loose, mushy stool (Diary-recorded stool consistency of 6 on the Bristol Stool Form Scale (BSFS or 4 on the modified Bristol Stool Form Scale for Children [mBSFSC]) or any watery stool (Diary-recorded stool consistency of 7 on the BSFS or 5 on the mBSFS-C) with any SBM that occurred in the absence of laxative use on the calendar day of the BM or the calendar day before the BM during each 7-day (week) period before the randomization day and up to the day of randomization;
20. ≥ 3 CSBMs per week for either week of the 2-week baseline diary assessment immediately preceding the randomization visit;
21. > 6 SBMs per week for either week of the 2-week baseline diary assessment immediately preceding the randomization visit;
22. Patient reports worst abdominal pain intensity (WAPI) scores in the 2-week baseline diary that meet either of the following:

    1. WAPI score of 0 on the 11-point Numeric Rating Scale or Wong-Baker Faces® Pain Rating Scale for more than two days during each week of the 2-week baseline diary period.
    2. An average WAPI < 3 for either of the two weeks of the baseline diary;
23. Completion of < 5 of the 7 required daily diary entries in each week of the 2-week baseline diary assessment immediately preceding the randomization visit;
24. Use of rescue medication (Dulcolax®, bisacodyl) for more than 2 days during either of the two weeks of the 2-week baseline diary assessment immediately preceding the randomization visit.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 218 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Bausch Site 178, Saraland, Alabama
  - Bausch Site 176, Scottsdale, Arizona
  - Bausch Site 160, Corona, California
  - Bausch Site 147, Garden Grove, California
  - Bausch Site 142, Los Angeles, California
  - Bausch Site 143, Ventura, California
  - Bausch Site 175, Aurora, Colorado
  - Bausch Site 197, Washington D.C., District of Columbia
  - Bausch Site 135, Doral, Florida
  - Bausch Site 190, Hialeah, Florida
  - Bausch Site 150, Miami, Florida
  - Bausch Site 130, Miami, Florida
  - Bausch Site 165, Miami, Florida
  - Bausch Site 110, Tampa, Florida
  - Bausch Site 174, Atlanta, Georgia
  - Bausch Site 132, Atlanta, Georgia
  - Bausch Site 148, Stockbridge, Georgia
  - Bausch Site 115, Evansville, Indiana
  - Bausch Site 139, Sioux City, Iowa
  - Bausch Site 192, Bowling Green, Kentucky
  - Bausch Site 172, Covington, Louisiana
  - Bausch Site 180, Crowley, Louisiana
  - Bausch Site 112, Lafayette, Louisiana
  - Bausch Site 220, Omaha, Nebraska
  - Bausch Site 145, Akron, Ohio
  - Bausch Site 194, Cleveland, Ohio
  - Bausch Site 111, Knoxville, Tennessee
  - Bausch Site 195, Austin, Texas
  - Bausch Site 225, Cedar Park, Texas
  - Bausch Site 173, Dallas, Texas
  - Bausch Site 193, Houston, Texas
  - Bausch Site 170, Houston, Texas
  - Bausch Site 140, San Antonio, Texas
  - Bausch Site 120, Newport News, Virginia
  - Bausch Site 146, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.0 mg Plecanatide - Group B: Plecanatide 1.0 mg Taken orally daily for 4 weeks Group B: 12 to18 years old
- 2.0 mg Plecanatide: Plecanatide 2.0 mg Taken orally daily for 4 weeks Group B: 12 to < 18 years old
  Plecanatide: Taken orally daily for 4 weeks
- Matching Placebo - Group B: Matching placebo tablets orally daily for 4 weeks Group B - 12 to 18 years old
Period: Overall Study
Arm/Group | 0.5 mg Plecanatide | 1.0 mg Plecanatide - Group A | Matching Placebo - Group A | 1.0 mg Plecanatide - Group B | 2.0 mg Plecanatide | 3.0 mg Plecanatide | Matching Placebo - Group B
Started | 30 | 29 | 29 | 34 | 32 | 32 | 32
Completed | 29 | 26 | 28 | 34 | 27 | 31 | 29
Not Completed | 1 | 3 | 1 | 0 | 5 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 2 | 0 | 0
Not completed — Participant moved and was unable to complete study | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Non-Compliance with eDiary | 1 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Non-Compliance with Study Drug | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) includes all randomized and treated subjects who have the baseline assessment and at least one post randomization assessment of the primary efficacy measure of weekly SBM frequency.
Groups:
- 1.0 mg Plecanatide - Group B: Plecanatide 1.0 mg Taken orally daily for 4 weeks Group B: 12 to 18 years old
- 2.0 mg Plecanatide: Plecanatide 2.0 mg Taken orally daily for 4 weeks Group B: 12 to < 18 years old
- Total: Total of all reporting groups
Arm/Group | 0.5 mg Plecanatide | 1.0 mg Plecanatide - Group A | Matching Placebo - Group A | 1.0 mg Plecanatide - Group B | 2.0 mg Plecanatide | 3.0 mg Plecanatide | Matching Placebo - Group B | Total
Number analyzed (Participants) | 30 | 29 | 29 | 34 | 32 | 32 | 32 | 218
Age, Customized [Count of Participants; unit: Participants]
  Age Group: Group A: Age 6 to 11 | 30 | 29 | 29 | 0 | 0 | 0 | 0 | 88
  Age Group: Group B: Age 12 to <18 | 0 | 0 | 0 | 34 | 32 | 32 | 32 | 130
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 15 | 20 | 20 | 20 | 20 | 126
  Male | 14 | 14 | 14 | 14 | 12 | 12 | 12 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 4 | 2 | 5 | 6 | 6 | 2 | 2 | 27
  White | 26 | 27 | 22 | 28 | 25 | 30 | 30 | 188
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 27 | 23 | 25 | 24 | 27 | 28 | 177
  Not Hispanic or Latino | 7 | 2 | 6 | 9 | 8 | 5 | 4 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 29 | 29 | 34 | 32 | 32 | 32 | 218
Height at Screening (m) [Mean (Standard Deviation); unit: meters] | 1.37 (0.136) | 1.36 (0.135) | 1.38 (0.131) | 1.63 (0.091) | 1.60 (0.097) | 1.58 (0.079) | 1.63 (0.086) | 1.51 (0.159)
Weight at Screening [Mean (Standard Deviation); unit: kilograms] | 37.53 (11.980) | 39.55 (15.118) | 38.79 (17.070) | 66.35 (22.402) | 60.72 (14.050) | 58.21 (16.223) | 63.60 (16.62) | 52.73 (20.231)
BMI at Screening [Mean (Standard Deviation); unit: kg/m^2] | 19.82 (4.961) | 20.87 (6.678) | 19.64 (5.590) | 24.85 (7.129) | 23.66 (4.460) | 23.26 (6.230) | 23.74 (4.867) | 22.385 (6.035)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Spontaneous Bowel Movement (SBM) Frequency Over the 4 Week Treatment Period Compared to Placebo and Across Treatment Groups
Description: Weekly SBM rate computed for each week
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: Number of SBMs per week
Groups:
- Experimental: 0.5 mg plecanatide: Plecanatide 0.5 mg Taken orally once daily for 4 weeks Group A: 6 to 11 years old
- Experimental: 1.0 mg plecanatide - Group A: Plecanatide 1.0 mg Taken orally daily for 4 weeks Group A: 6 to 11 years old
- Experimental: 1.0 mg plecanatide - Group B: Plecanatide 1.0 mg Taken orally daily for 4 weeks Group B: 12 to18 years old
- Experimental: 2.0 mg plecanatide: Plecanatide 2.0 mg Taken orally daily for 4 weeks Group B: 12 to < 18 years old
- Experimental: 3.0 mg plecanatide: Plecanatide 3.0 mg Taken orally daily for 4 weeks Group B: 12 to < 18 years old
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | Experimental: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching Placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Number of SBMs per week | 0.6 (2.24) [-0.86 to 0.90] | 0.8 (1.75) [-0.65 to 1.17] | 0.6 (1.53) | 1.0 (2.08) [-0.06 to 1.87] | 1.1 (2.20) [0.05 to 2.01] | .70 (2.45) [-0.28 to 1.67] | -0.2 (1.95)

2. Secondary Outcome: Change From Baseline in Frequency of Abdominal Pain and Abdominal Discomfort Over the 4-week Treatment Period Compared to Placebo and Across Treatment Groups..
Description: Weekly frequency was calculated as the number of abdominal pain episodes and abdominal discomfort episodes per week, based on daily diary entries. Baseline was the average weekly frequency during the 2-week baseline assessment period. Values shown are mean change from baseline (SD).
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: Episodes per week
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | ExperimentaL: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Episodes per week
  Frequency of Abdominal Pain | -2.7 (2.27) | -2.2 (2.38) | -1.4 (2.47) | -1.3 (1.49) | -1.6 (2.34) | -1.4 (2.26) | -1.6 (2.56)
  Frequency of Abdominal Discomfort | -2.5 (2.18) | -2.1 (2.35) | -1.3 (2.44) | -0.9 (1.59) | -1.5 (2.22) | -1.1 (2.03) | -1.3 (2.43)

3. Secondary Outcome: Change From Baseline in Severity of Abdominal Pain and Abdominal Discomfort Over the 4-week Treatment Period Compared to Placebo and Across Treatment Groups..
Description: Severity of abdominal pain and abdominal discomfort was recorded daily using an electronic diary on a 0-10 numeric rating scale (0 = no pain/discomfort; 10 = worst possible). Weekly averages were calculated; baseline was the average score during the 2-week baseline period. Values shown are mean change from baseline.
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: Severity score (0-10 scale)
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | ExperimentaL: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Severity score (0-10 scale)
  Severity of Abdominal Pain | -3.3 (3.07) [-1.39 to 0.88] | -2.3 (2.72) [-0.62 to 1.69] | -2.3 (2.33) | -2.2 (2.37) [-1.09 to 0.77] | -2.8 (2.19) [-1.70 to 0.2] | -2.56 (2.27) [-1.22 to 0.67] | -2 (2.36)
  Severity of Abdominal Discomfort | -3.4 (2.97) [-2.24 to 0.18] | -2.4 (2.83) [-1.25 to 1.22] | -2.40 (2.51) | -1.9 (2.58) [-1.00 to 1.01] | -3.0 (2.23) [-1.97 to 0.10] | -2.5 (2.36) [-1.47 to 0.58] | -2.0 (2.46)

4. Secondary Outcome: Change From Baseline in Frequency of Complete Spontaneous Bowel Movements (CSBM)
Description: Weekly frequency of complete spontaneous bowel movements (CSBMs) was calculated based on daily diary entries. Baseline was the average weekly frequency during the 2-week baseline period. Values shown are mean change from baseline (SD) at end of 4 weeks of study.
Time Frame: Baseline to Week 6
Measure: Mean (Standard Deviation); unit: Change in Number of CSBMs per week
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | Experimental: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Change in Number of CSBMs per week | 0.7 (1.73) | 0.2 (0.75) | 0.2 (0.91) | 0.4 (0.85) | 0.1 (1.07) | 0.7 (1.79) | -0.1 (0.47)

5. Secondary Outcome: Change From Baseline in Frequency of Bowel Movements (BM)
Description: Weekly frequency of bowel movements (BMs) was calculated based on daily diary entries. Baseline was the average weekly frequency during the 2-week baseline period. Values shown are mean change from baseline (SD).
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: Number of BMs per week
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | Experimental: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Number of BMs per week | 0.5 (2.24) | 0.8 (1.7) | 0.6 (1.52) | 0.8 (2.06) | 1.0 (2.23) | 0.8 (2.263) | 0 (2.05)

6. Secondary Outcome: Time to First Bowl Movement (in Days)
Description: This outcome was analyzed as a time-to-event variable (time to first complete spontaneous bowel movement), and confidence intervals were estimated using Kaplan-Meier methods.
Time Frame: Day 1 to first BM during Treatment Period
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | Experimental: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching Placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Days | 4.1 [1.13 to 11.43] | 2.58 [1.56 to 6.21] | 5.35 [2.35 to NA] — The upper confidence limit could not be estimated because the time-to-event distribution did not contain a sufficient number of events beyond the median to support calculation of the upper confidence interval. | 1.68 [0.99 to 5.23] | 2.05 [0.86 to 6.25] | 2.57 [0.89 to 8.15] | 2.69 [1.35 to 5.28]

7. Secondary Outcome: Change From Baseline in Stool Consistency (Based on Bristol Stool Form Scale, BSFS or Modified Bristol Stool Form Scale for Children, mBSFS-C)
Description: Weekly stool consistency scores based on BSFS (≥12 years) or mBSFS-C (6-11 years). BSFS Scale is a 7 point scale, from Type 1 (Hard to pass) to Type 7 (entirely liquid). mBSFS-C is a 5 point scale, from Type 1 (hard to pass) to Type 5 (watery, no solid pieces).
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: Score (BSFS or mBSFS-C)
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | Experimental: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Score (BSFS or mBSFS-C) | 1.2 (1.12) | 0.8 (1.18) | 1.2 (0.72) | 1.1 (1.24) | 1.4 (1.5) | 1.9 (1.35) | 0.7 (0.96)

8. Secondary Outcome: Use of Rescue Medication
Description: Number of rescue medication tablets (Dulcolax® 5 mg) used during the 4-week treatment period. Subjects were instructed to use rescue medication only if ≥72 hours had passed since last bowel movement.
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: Number of Tablets
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | Experimental: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching Placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Number of Tablets | 1.3 (3.6) | 0.7 (3.22) | 0.4 (1.18) | 2.4 (8.73) | 0.2 (0.59) | 1.6 (5.02) | 2.4 (6.68)

9. Secondary Outcome: Change From Baseline in Frequency of Fecal Incontinence
Description: Weekly fecal incontinence episodes recorded in daily diary.
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: Number of episodes per week
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | Experimental: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching Placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Number of episodes per week | 0.3 (2.10) | 1.9 (4.36) | 1.1 (3.04) | 0.9 (2.58) | 2.3 (5.33) | 1.0 (2.73) | 1.3 (3.29)

10. Secondary Outcome: Change From Baseline in Severity of Defecation Pain
Description: Severity of abdominal pain scored daily on a 0-10 numeric rating scale (0 = no pain, 10 = worst possible pain). Weekly averages were calculated from daily scores.
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: Severity Score 0-10 scale
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | Experimental: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching Placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Severity Score 0-10 scale | -2.4 (3.13) | -2.6 (3.16) | -2.6 (3.62) | -2.3 (2.98) | -2.5 (2.17) | -1.8 (2.7) | -1.6 (2.83)

11. Secondary Outcome: Change From Baseline in Frequency of Pain With Defecation
Description: Pain with defecation was recorded in daily diaries as the number of episodes per week. Results represent the mean change from baseline in weekly frequency.
Time Frame: Baseline to Week 4
Population: All randomized participants who received at least one dose of study drug and had both baseline and post-baseline pain frequency assessments.
Measure: Mean (Standard Deviation); unit: Change in Episodes per week
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | Experimental: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching Placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Change in Episodes per week | -0.3 (2.64) | -0.8 (2.97) | -0.3 (2.91) | 0.4 (2.33) | -0.5 (2.29) | -0.8 (2.55) | -0.7 (2.58)

12. Secondary Outcome: Change From Baseline in Frequency of Large Diameter Stools
Description: Weekly frequency of large diameter stools recorded in daily diary.
Time Frame: Baseline to Week 4
Measure: Mean (Standard Deviation); unit: Number of episodes per week
Arm/Group | Experimental: 0.5 mg plecanatide | Experimental: 1.0 mg plecanatide - Group A | Matching placebo - Group A | Experimental: 1.0 mg plecanatide - Group B | Experimental: 2.0 mg plecanatide | Experimental: 3.0 mg plecanatide | Matching Placebo - Group B
Number analyzed (Participants) | 30 | 28 | 29 | 34 | 32 | 32 | 32
Number of episodes per week | 0 (.28) | 0 (0.48) | 0.1 (0.57) | 0.0 (0.61) | -0.1 (0.49) | 0.0 (0.40) | 0.1 (0.67)

ADVERSE EVENTS:
Time Frame: From consent signature until end of study participation, up to 10 weeks. This includes screening, 4-week treatment, and 2-week follow-up periods.
Description: Adverse events were coded using MedDRA Version 24.1. All AEs were collected from consent through final study visit, regardless of relationship to study drug.
  GI symptoms (e.g., abdominal pain, discomfort, defecation pain) were captured via daily electronic diaries and not separately reported as AEs unless considered bothersome by the subject.
  Missing severity or relationship values were imputed as "Severe" and "Reasonable Possibility," respectively.
Arm/Group | Experimental: 0.5 mg Plecanatide | Experimental: 1.0 mg Plecanatide - Group A | Matching Placebo - Group A | Experimental: 1.0 mg Plecanatide - Group B | Experimental: 2.0 mg Plecanatide | Experimental: 3.0 mg Plecanatide | Matching Placebo - Group B
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29 | 0/29 | 0/34 | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/29 | 0/34 | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 2/30 | 5/29 | 1/29 | 7/34 | 3/32 | 3/32 | 2/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: 0.5 mg Plecanatide (N=30) | Experimental: 1.0 mg Plecanatide - Group A (N=29) | Matching Placebo - Group A (N=29) | Experimental: 1.0 mg Plecanatide - Group B (N=34) | Experimental: 2.0 mg Plecanatide (N=32) | Experimental: 3.0 mg Plecanatide (N=32) | Matching Placebo - Group B (N=32)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) — Mild
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Mild
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Mild
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Mild
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Mild
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT03596905/Prot_SAP_000.pdf